CLINICAL TRIAL: NCT00744354
Title: A Phase 1 Dose Escalation Study of Bortezomib (Velcade®), Pegylated Liposomal Doxorubicin (Doxil®), and Vorinostat (Suberoylanilide Hydromaxic Acid, Saha, Zolinzatm) in Patients With Relapse/Refractory Multiple Myeloma
Brief Title: Vorinostat, Bortezomib, and Doxorubicin Hydrochloride Liposome in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs unavailable- study terminated 1/2/18
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Millennium Pharmaceuticals, Inc. (Industry); Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0715; 08-1073 (Other: Office of Human Research Ethics)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; liposomal doxorubicin; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Randomized Open Label Single Arm (Experimental): Phase 1 dose escalation trial of vorinostat in combination with bortezomib and pegylated liposomal doxorubicin hydrochloride.
  Interventions: Drug: bortezomib; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vorinostat

INTERVENTIONS:
Drug: bortezomib — Intravenous Push 1.3 mg/m2 Days 1, 4, 8, and 11
  Other Names: Velcade
Drug: pegylated liposomal doxorubicin hydrochloride — Intravenous infusion, 30mg/m2, Day 4, each cycle
  Other Names: Doxil
Drug: vorinostat — Oral, 300mg, Days 1, 2, 4, 5, 8, 9, 11, 12, every cycle.
  Other Names: Zolinza

SUMMARY:
RATIONALE: Vorinostat and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bortezomib may also stop the growth of multiple myeloma by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving doxorubicin hydrochloride liposome together with vorinostat and bortezomib may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat and to see how well it works when given together with bortezomib and doxorubicin hydrochloride liposome in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of vorinostat when added to the standard regimen of bortezomib and pegylated liposomal doxorubicin hydrochloride in patients with relapsed or refractory multiple myeloma.
* To identify the dose-limiting toxicities of this regimen in these patients.

Secondary

* To gain preliminary evidence of antitumor activity of this regimen in these patients.
* To assess the degree of proteasome inhibition achieved with this regimen in these patients.
* To evaluate the accumulation of acetylated alpha-tubulin after treatment with vorinostat.
* To evaluate overall survival, time to progression, and progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose escalation study of vorinostat.

Patients receive oral vorinostat once daily on days 1,2; 4,5; 8, 9; 11, 12; bortezomib IV on days 1, 4, 8, and 11, and pegylated liposomal doxorubicin hydrochloride IV on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for proteasome inhibition assays and acetylated alpha-tubulin studies.

After completion of study treatment, patients are followed at 1 and 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Relapsed or refractory disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1.0 x 10^9/L (no granulocyte growth factor support, e.g., G-CSF or GM-CSF allowed)
* Platelet count ≥ 100 x 10^9/L (erythropoietin allowed, no platelet or RBC transfusion within the past 2 weeks)
* Hemoglobin ≥ 8 g/dL (erythropoietin allowed, no platelet or RBC transfusion within the past 2 weeks)
* Creatinine clearance ≥ 30 mL/min
* AST or ALT ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* LVEF ≥ 45% by MUGA or ECHO
* Symptomatic neuropathy < grade 2
* No known history of HIV
* No active or serious infection, medical or psychiatric illness that would preclude study participation
* No active hepatitis B or C infection
* No other prior or concurrent malignancy except for adequately treated basal cell or squamous cell carcinoma of the skin, in situ malignancy, low-risk prostate cancer after curative therapy, or other cancer for which the patient has been disease-free for ≥ 3 years
* No history of hypersensitivity reaction to bortezomib or any of its components (boron, mannitol), vorinostat, doxorubicin hydrochloride, or any of the components of PLD
* No serum potassium ≤ 3.0 or serum magnesium ≤ 1.6 that cannot be corrected with supplementation are excluded
* Patients must have adequate cardiovascular function, defined by all of the following:

  * No EKG evidence of active, clinically significant conduction system abnormalities
  * No EKG evidence of QTc prolongation > grade 2
* NOTE: Any EKG abnormality at screening has to be documented by the investigator as not medically significant.

PRIOR CONCURRENT THERAPY:

* No limit to number of prior treatment regimens
* At least 30 days since prior therapy and recovered
* At least 3 months since prior autologous stem cell transplantation and recovered
* Prior allogeneic stem cell or bone marrow transplantation allowed provided the following criteria are met:

  * More than 1 year since transplantation
  * No longer receiving immunosuppressive therapy or treatment for graft-versus-host disease (GVHD) prophylaxis
  * No active GVHD
  * No active, uncontrolled infections
* No major surgery within the past 3 weeks
* No prior anthracycline dose > 360 mg/m^2 for doxorubicin hydrochloride (including pegylated liposomal doxorubicin hydrochloride [PLD]) or 720 mg/m^2 for epirubicin hydrochloride
* No prior or concurrent histone deacetylase inhibitor (e.g., valproic acid)
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) during course 1
* No other concurrent investigational or anticancer agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat | 4 years

SECONDARY OUTCOMES:
Overall response rate | 5 years
Duration of response | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brandi Reeves, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- See also: Web address for UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org